CLINICAL TRIAL: NCT00930644
Title: A Long-Term, Open-Label Study With Teduglutide for Subjects With Parenteral Nutrition Dependent Short Bowel Syndrome
Brief Title: Open-Label Study of Teduglutide for Subjects With PN-Dependent Short Bowel Syndrome (SBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Nycomed Germany GmbH (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0600-021; 2009-011679-65 (EudraCT Number)
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Short Bowel Syndrome
Keywords: short bowel syndrome; parenteral nutrition; PN; HPN; TPN; SBS
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- teduglutide (Experimental): 0.05 mg/kg/day
  Interventions: Drug: teduglutide

INTERVENTIONS:
Drug: teduglutide — 0.05 mg/kg/day subcutaneously taken once per day for 24 months
  Other Names: Gattex

SUMMARY:
This study is a 2-year open label extension study to collect long term efficacy and safety data from patients who have completed the 24-weeks of study drug dosing in CL0600-020.

DETAILED DESCRIPTION:
Some people with SBS need to infuse parenteral nutrition (PN) in order to live. Although PN can save lives, it can lead to some serious side effects such as infection or liver damage. The risk for those effects increases the longer people are on PN.

Teduglutide is an investigative medicine being evaluated as a possible treatment for people with PN-dependent SBS. Teduglutide is similar to a protein the body makes. When people have SBS, their bodies do not make enough of the protein and they have trouble getting nutrients and fluids from the food they eat and drink. We want to see if teduglutide can help decrease the amount of PN needed because the body is doing a better job of taking up what it eats and drinks. We also want to find out how safe teduglutide is and record any side effects.

ELIGIBILITY:
Inclusion Criteria:

* must have completed 24 weeks of dosing of the CL0600-020 study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-09-21 (Actual); Primary Completion 2013-01-24 (Actual); Study Completion 2013-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (6):
  - Scripps Clinic & Research Foundation, La Jolla, California
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennslyvania, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (3):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hôpital Beaujon, Clichy
  - Hopital de l'Archet 2, Nice
- Germany (2):
  - Universitaetsklinikum Tuebingen Medizinische Klinik I, Tübingen, Baden-Wurttemberg
  - Med. Klinik m.S. Hepatologie und Gastroenterologie, Berlin, State of Berlin
- Azienda Universitaria Policlinico Federico II, Napoli, Italy
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny im. M. Pirogowa, Pracownia Leczenia Zywieniowego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Klinika Chirurgii Ogolnej i Transplantacyjnej, Lublin
  - Pracownia Żywienia Klinicznego, Olsztyn
  - Samodzielny Publiczny Szpital Kliniczny-Im.prof W.Orłowskiego CMKP, Warsaw
- Spain (2):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - St. Marks Hospital, Harrow
  - University College London Hospital, London

REFERENCES:
- [Background] Jeppesen PB, Sanguinetti EL, Buchman A, Howard L, Scolapio JS, Ziegler TR, Gregory J, Tappenden KA, Holst J, Mortensen PB. Teduglutide (ALX-0600), a dipeptidyl peptidase IV resistant glucagon-like peptide 2 analogue, improves intestinal function in short bowel syndrome patients. Gut. 2005 Sep;54(9):1224-31. doi: 10.1136/gut.2004.061440. PMID 16099790
- [Derived] Pape UF, Iyer KR, Jeppesen PB, Kunecki M, Pironi L, Schneider SM, Seidner DL, Lee HM, Caminis J. Teduglutide for the treatment of adults with intestinal failure associated with short bowel syndrome: pooled safety data from four clinical trials. Therap Adv Gastroenterol. 2020 Apr 20;13:1756284820905766. doi: 10.1177/1756284820905766. eCollection 2020. PMID 32341691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met any of the following could be enrolled: Completed 24 weeks of treatment in Study CL0600-020; based on PI and sponsor decision, subjects who were required to stop treatment prematurely due to a non drug related AE; or successfully completed Stage I (optimization/stabilization) in Study CL0600-020 after ~86 subjects were randomized
Groups:
- Teduglutide 0.05 mg/kg/Day: teduglutide: 0.05 mg/kg/day subcutaneously taken once per day for 24 months
Period: Overall Study
Arm/Group | Teduglutide 0.05 mg/kg/Day
Started | 88
Completed | 65
Not Completed | 23
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Death | 1
Not completed — Adverse Event | 16

BASELINE CHARACTERISTICS:
Arm/Group | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 73
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 41
Years since start of PN/IV dependecy [Mean (Standard Deviation); unit: years] | 6.41 (6.272)
Prescribed weekly PN/IV volume [Mean (Standard Deviation); unit: Liters] | 12.07 (7.56)
Prescribed weekly number of days on PN/IV [Mean (Standard Deviation); unit: days] | 5.6 (1.68)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in PN/IV Volume by Visit
Description: The mean change from baseline in weekly PN.IV volume in percent change is shown by visit.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- NT/TED: No treatment in CL0600-020 trial and teduglutide 0.05 mg/kg/day subcutaneously taken once per day for 24 months in CL0600-021 trial
- PBO/TED: Placebo in CL0600-020 trial and teduglutide 0.05 mg/kg/day subcutaneously taken once per day for 24 months in CL0600-021 trial
- TED/TED: 0.05 mg/kg/day subcutaneously taken once per day for 6 months CL0600-020 trial and teduglutide 0.05 mg/kg/day subcutaneously taken once per day for 24 months in CL0600-021 trial
Arm/Group | NT/TED | PBO/TED | TED/TED
Number analyzed (Participants) | 12 | 39 | 37
percent change
  Month 1 | -5.35 (11.287) | -6.44 (11.241) | -40.65 (21.546)
  Month 2 | -12.88 (22.789) | -10.27 (14.027) | -44.24 (21.823)
  Month 3 | -10.83 (47.396) | -14.18 (16.440) | -45.80 (22.681)
  Month 6 | -24.13 (17.496) | -16.48 (20.979) | -34.70 (55.319)
  Month 9 | -25.35 (17.855) | -20.95 (27.500) | -37.91 (57.460)
  Month 12 | -23.33 (20.296) | -22.00 (33.858) | -51.33 (28.299)
  Month 15 | -31.62 (25.901) | -18.89 (33.165) | -54.24 (27.871)
  Month 18 | -35.11 (35.545) | -24.18 (32.183) | -63.01 (26.587)
  Month 21 | -39.40 (36.504) | -27.67 (33.064) | -64.99 (27.920)
  Month 24 | -39.40 (36.504) | -28.33 (35.169) | -65.61 (33.606)

2. Primary Outcome: Absolute Change in PN/IV Volume by Visit
Description: The mean change from baseline in weekly PN.IV volume in Liters is shown by visit.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NT/TED | PBO/TED | TED/TED
Number analyzed (Participants) | 12 | 39 | 37
Liters
  Month 1 | -1.05 (1.315) | -0.95 (1.938) | -5.28 (3.819)
  Month 2 | -1.88 (2.057) | -1.38 (2.228) | -5.62 (3.873)
  Month 3 | -2.55 (3.123) | -1.65 (2.456) | -5.72 (3.771)
  Month 6 | -3.85 (2.761) | -1.90 (3.309) | -5.20 (4.650)
  Month 9 | -3.69 (2.916) | -2.61 (4.071) | -5.59 (4.899)
  Month 12 | -2.90 (2.762) | -2.72 (4.310) | -6.36 (4.633)
  Month 15 | -3.58 (2.811) | -2.48 (4.398) | -6.37 (4.261)
  Month 18 | -3.63 (2.834) | -2.90 (4.394) | -6.99 (4.048)
  Month 21 | -4.01 (2.910) | -3.00 (3.571) | -7.34 (4.412)
  Month 24 | -4.01 (2.910) | -3.11 (3.880) | -7.55 (4.930)

3. Secondary Outcome: Number of Subjects Achieving PN/IV Reduction
Description: The number of subjects who achieve at least 1-, 2-, and 3-day reductions in PN/IV per Week.
Time Frame: 24 Months or Last Dosing Visit
Measure: Number; unit: participants
Arm/Group | NT/TED | PBO/TED | TED/TED
Number analyzed (Participants) | 12 | 39 | 37
participants
  Achieving >= 1 Day of PN/IV Reduction | 3 | 14 | 21
  Achieving >= 2 Day of PN/IV Reduction | 2 | 7 | 18
  Achieving >= 3 Day of PN/IV Reduction | 2 | 5 | 18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject from the time informed consent was signed to the end of the study. The most commonly reported treatment emergent adverse events (>= 3% grouped at PT level) are listed.
Description: Adverse events monitoring was performed through investigator assessment and safety laboratory testing at each visit.
Groups:
- NT,PBO/TED: No treatment or placebo in CL0600-020 trial and teduglutide 0.05 mg/kg/day subcutaneously taken once per day for 24 months in CL0600-021 trial
Arm/Group | NT,PBO/TED | TED/TED
Serious Adverse Events (participants affected / at risk) | 32/51 | 24/37
Other Adverse Events (participants affected / at risk) | 49/51 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT,PBO/TED (N=51) | TED/TED (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Crohns disease (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fecal volume increased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (7) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 3 (5) | 5 (7)
Catheter bacteraemia (Infections and infestations) | 4 (7) | 0 (0)
Catheter sepsis (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4)
Catheter site infection (Infections and infestations) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2)
Hepatic cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Chemical burn of the eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device breakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Gamma glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Nervous system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena caval stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT,PBO/TED (N=51) | TED/TED (N=37)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 5 (10) | 3 (5)
Gastrointestinal Disorders (Gastrointestinal disorders) | 34 (148) | 20 (68) — Includes abdominal pain, nausea, abdominal distension, diarrhea, flatulence, vomiting, abdominal pain upper, dyspepsia, abdominal discomfort, constipation, faecal volume increased, intestinal obstruction, abdominal pain lower, and others.
General Disorders, and Administration Site Conditions (General disorders) | 27 (100) | 15 (40)
Hepatobiliary Disorders (Hepatobiliary disorders) | 8 (10) | 2 (2)
Infections and Infestations (Infections and infestations) | 31 (97) | 26 (62)
Injury, Poisoning, and Procedural Complications (Injury, poisoning and procedural complications) | 19 (39) | 13 (39)
Investigations (Investigations) | 22 (62) | 19 (31)
Metabolism and Nutrition Disorder (Metabolism and nutrition disorders) | 14 (44) | 14 (33)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 11 (37) | 13 (23)
Nervous System Disorders (Nervous system disorders) | 10 (60) | 10 (18)
Psychiatric Disorders (Psychiatric disorders) | 8 (11) | 2 (2)
Renal and Urinary Disorders (Renal and urinary disorders) | 6 (17) | 4 (17)
Respiratory, Thoracic, and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 10 (20) | 7 (9)
Vascular Disorder (Vascular disorders) | 14 (18) | 6 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of NPS Pharmaceuticals agreements with its investigators may vary. However, NPS does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e. data from all sites) in the clinical trial.